CLINICAL TRIAL: NCT01792063
Title: A Randomized Clinical Trial on the Efficiency, Hemodynamic Effects and Patient Comfort of Two Different Preparations of Sevoflurane After Vital Capacity Rapid Inhalation Induction
Brief Title: Two Different Preparations of Sevoflurane in Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Assoc.Prof, Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 43430
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Coughing on Induction; Vapors; Inhalation
MeSH Terms: conditions — Respiratory Aspiration | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane A (Active Comparator): Generic sevoflurane
  Interventions: Drug: Sevoflurane
- Sevoflurane B (Active Comparator): Orginal sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane
  Other Names: Sevorane, Abbott Laboratories
  Arms: Sevoflurane A
Drug: Sevoflurane
  Other Names: Sojourn, Adeka IS A.S
  Arms: Sevoflurane B

SUMMARY:
In our study we aim to study the effects of two preparations of Sevoflurane in vital capacity rapid inhalation induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal surgery

Exclusion Criteria:

* Patients with any cardiovascular or respiratory disease, usage of any kind of sedative drug, expected airway difficulty and obese patients (BMI>35) will be excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
effect of different preparations of sevoflurane on Induction on hypnosis time | 1 hour
  Induction for anesthesia will be achieved with sevoflurane A and Sevoflurane B in total of 100 randomized (American Society of Anesthesiology status I-II) patients undergoing abdominal surgery. During the induction patients will be asked to breath as deep as possible and then hold their breaths to the point where they cannot anymore and flexing their right arm. Occurrence of hypnosis will be confirmed with both the loss of eyelash-reflex and failing of flexed-holding arm. Time and number of breaths needed for the loss of consciousness will be noted. Existence of hiccup, cough, increase in secretions, and refusal of the mask by the patient will be reported if any. All patients will be extubated and released to the ward after they are questioned about any discomfort or issue they want to report to anesthesiologist

SECONDARY OUTCOMES:
effect of different sevoflurane preparations on hemodynamics | 1 hour
  After the induction and occurrence of hypnosis, Systemic arterial pressure (SAP) values will be noted. Tracheal intubation will be performed and post-intubation SAP values will be noted. The SAP values will noted in the 5th minute of the induction.

CONTACTS AND LOCATIONS:
Locations (1):
- Cerrahpasa Medical Faculty Anesthesiology and Reanimation Department, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Baker MT. Sevoflurane: are there differences in products? Anesth Analg. 2007 Jun;104(6):1447-51, table of contents. doi: 10.1213/01.ane.0000263031.96011.36. PMID 17513639